CLINICAL TRIAL: NCT01763190
Title: An Open-label Pharmacokinetic and Tolerability Study of SAR302503 Given as a Single 300 mg Dose in Subjects With Mild, Moderate and Severe Renal Impairment, and in Matched Subjects With Normal Renal Function
Brief Title: Open Label Pharmacokinetic Study of SAR302503 in Subjects With Renal Impairment
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: POP13449; U1111-1115-8416 (Other: UTN)
Record Dates: First submitted 2013-01-04; First posted 2013-01-08 (Estimated); Last update posted 2025-03-05 (Actual); Status verified 2015-05

CONDITIONS: Renal Impairment
MeSH Terms: conditions — Renal Insufficiency | interventions — fedratinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- SAR302503 (Experimental): single treatment of 300 mg oral dose of SAR302503
  Interventions: Drug: SAR302503

INTERVENTIONS:
Drug: SAR302503 — Pharmaceutical form:capsule
  Route of administration: oral

SUMMARY:
Primary Objective:

To study the effect of mild, moderate and severe renal impairment on the pharmacokinetics of SAR302503.

Secondary Objective:

To assess the tolerability of SAR302503 given as a single 300 mg dose in subjects with mild, moderate and severe renal impairment and in matched subjects with normal renal function.

DETAILED DESCRIPTION:
study duration = 17 to 35 days

ELIGIBILITY:
Inclusion criteria :

* Male or female subjects, between 18 and 75 years of age, inclusive.
* For subjects between ages 75 to 79 with the approval from sponsor's medical monitor.
* Body weight between 50.0 and 115.0 kg, inclusive if male, and between 40.0 and 100.0 kg, inclusive if female, body mass index between 18.0 and 34.9 kg/m2, inclusive.
* Stable chronic renal impairment, as defined by Cockcroft-Gault formula;
* Laboratory parameters within the acceptable range for subjects with renal impairment.
* Using a double contraception method.

Exclusion criteria:

* Uncontrolled clinically relevant cardiovascular, pulmonary, gastrointestinal, metabolic,hematological, neurological, psychiatric, systemic, ocular, gynecologic (if female), or infectious disease, or signs of acute illness
* Active hepatitis, hepatic insufficiency
* Acute renal failure (de novo or superimposed to preexisting chronic renal impairment), nephrotic syndrome
* History of or current hematuria of urologic origin that limits the subject's participation in the study
* Subjects requiring dialysis during the study.
* Any significant change in chronic treatment medication within 14 days before inclusion.
* Concomitant treatment with or use of drugs or herbal agents known to be at least moderate inhibitors or inducers CYP3A4, sensitive or narrow therapeutic index substrate of CYP3A4.
* Concomitant treatment with gastric pH modifying agents (proton pump inhibitors and H2-blockers) is not allowed 7 days prior to and 6 hours after study drug treatment

The above information is not intended to contain all considerations relevant to a patient's potential participation in a clinical trial.

Ages: 18 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2012-11; Primary Completion 2013-07 (Actual); Study Completion 2013-07 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetic parameter: Cmax, AUClast and AUC | 12 days

SECONDARY OUTCOMES:
Pharmacokinetic parameters : unbound AUC, unbound Cmax, CL/F, Vss/F , t1/2z, t1/2eff, Rac, pred | 12 days
Safety parameters including Clinical tests | 16 days
Safety parameters including laboratory tests | 16 days
Safety parameters including ECG parameters | 16 days
Number of subjects with adverse events (AEs) | 16 days

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi
Locations (3):
- United States (3):
  - Investigational Site Number 840002, Orlando, Florida
  - Investigational Site Number 840003, Saint Paul, Minnesota
  - Investigational Site Number 840001, Knoxville, Tennessee